CLINICAL TRIAL: NCT06013657
Title: Surgical Resection for Hepatocellular Carcinoma: a Single-Center's One Decade of Experience
Brief Title: Surgical Resection for Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Ridho Ardhi Syaiful, Principal investigator, Dr Cipto Mangunkusumo General Hospital
Other Study IDs: DRCiptoMGH 19-11-1313
Record Dates: First submitted 2023-08-15; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Resectable Hepatocellular Carcinoma
Keywords: carcinoma,hepatocellular; liver neoplasms; hepatectomy; mortality; prognostic
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver resection: Patients undergoing liver resection due to hepatocellular carcinoma from 2010 to 2021 in RSCM, Jakarta, an academic tertiary-level national referral hospital in Indonesia.
  Interventions: Procedure: Liver Resection

INTERVENTIONS:
Procedure: Liver Resection — Resection of a part of the liver afflicted by hepatocellular carcinoma
  Other Names: Hepatectomy

SUMMARY:
Hepatocellular carcinoma is a type of liver cancer and is one of the leading causes of global cancer death. Surgical resection of the afflicted areas of the liver is one of the treatment methods for this condition. In this retrospective research, the investigators explore the outcomes of liver resection for hepatocellular carcinoma patients undergoing liver resection from 2010 to 2021 in Cipto Mangunkusumo General Hospital, Jakarta. The main outcome is mortality and the secondary outcomes are factors predicting mortality after resection.

DETAILED DESCRIPTION:
Study design This is a retrospective cohort study.

Treatment of Hepatocellular Carcinoma Patients in RSCM HCC patients are managed by a multidisciplinary team (MDT) consisting of hepatologists, radiologists, pathologists, radiation oncologists, surgeons, and other specialists related to the patient's condition. Confirmed HCC patients are discussed in a weekly MDT team meeting. The meeting assigned patients to treatment options according to the Barcelona Clinic Liver Center (BCLC) staging system, patient preference, and other clinical considerations. Resection is considered for patients at very early (BCLC 0) or early (BCLC A) HCC stages. This includes CP class A patients with a single tumor or less than three small (<3 cm) tumors. Patients assigned to surgical resection underwent either laparoscopic or open surgery. One to four segments of the liver were removed. Tissue samples were taken for further pathologic examination.

Ethical Clearance The ethics committee of The Faculty of Medicine, University of Indonesia, approved this study by giving an ethical clearance with protocol number 19-11-1313. Informed consent was taken from all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing liver resection in Cipto Mangunkusumo hospital due to a confirmed diagnosis of hepatocellular carcinoma from 2010 to 2021

Exclusion Criteria:

* Patients undergoing liver resection in other hospitals were excluded, even though diagnosis or further care is done in Cipto Mangunkusumo hospital
* Patients with other malignancies
* Patients undergoing other treatment methods for hepatocellular carcinoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study used a total population sampling of all patients undergoing liver resection in Cipto Mangunkusumo hospital due to a confirmed diagnosis of hepatocellular carcinoma from 2010 to 2021. Patients undergoing liver resection in other hospitals were excluded, even though diagnosis or further care is done in RSCM. In addition, patients with other malignancies or undergoing other treatment methods were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Mortality | Through study completion, an average of 3 years
  Mortality status of patients

SECONDARY OUTCOMES:
Age | Within one week before surgery
  Age in years
Sex | Within one week before surgery
  Male or Female
Etiology | Within one month before surgery
  Divided into hepatitis B, hepatitis C, and non-hepatitis in accordance with the laboratory results.
Child-Pugh classification | Within one month before surgery
  Divided into Chilld-Pugh A,B, and C using clinical (presence of encephalopathy or ascites) and laboratory (prothrombin time, albumin, and bilirubin levels) data.
BCLC Classification | Within one month before surgery
  Divided into Stages 0 and A to D using performance status, child-pugh classification, number and size (in cm) of the tumor.
AFP Levels | Within one month before surgery
  Divided into <400 and >=400
Number of tumors | Within one month before surgery
  Divided into single and multiple tumors according to imaging findings
Largest diameter of tumor | Within one month before surgery
  Measured in cm according to imaging
Surgery method | During surgery
  Laparoscopy or open surgery
Segments resected | During surgery
  1-4 segments
Cirrhosis | Within one month after surgery
  Presence of cirrhosis in histopathological findings
Edmondson's grading | Within one month after surgery
  Histopathological grading divided into 1 to 4
Tumor differentiation | Within one month after surgery
  Histopathological grading divided well, moderate, moderate to poor, and poor
Length of stay | An average of two weeks
  Measured in days from admission to discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
Raw data without the patients' identification in the form of an Excel sheet will be made available per private request via e-mail correspondence.